CLINICAL TRIAL: NCT06284239
Title: An Example of the Tell Me Game in Nursing History Teaching: Randomized Controlled Research
Brief Title: Using Games in Teaching Nursing History
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Tell Me Game
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Education Nursing

STUDY DESIGN:
Intervention Model Description: It refers to the intervention group in which the "Tell Me" game will be played.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed about the research. However, participants will not know which group they belong to. At the same time, the statistical analysis of the research will be carried out by an independent statistician. Thus, blinding of both the participant and the outcome assessor will be ensured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): For six weeks, theoretical training on the history of Nursing will be given by the researchers. Then, all the topics learned in the course will be repeated using question-answer and discussion methods, using questions prepared by the researchers, with the control group for four weeks. After this process, carried out by one of the researchers, is completed, the students will be given a nursing history knowledge test (posttest) and a nursing history teaching evaluation form and asked to fill it out.
- Interversion group (Experimental): For six weeks, theoretical training on the history of Nursing will be given by the researchers. Then, the intervention group will be played the tell-all game with game cards prepared by the researchers for four weeks. After this process, carried out by one of the researchers, is completed, the students will be given a nursing history knowledge test (posttest) and a nursing history teaching evaluation form and asked to fill it out.
  Interventions: Other: Tell me about the game.

INTERVENTIONS:
Other: Tell me about the game. — It is a game played with playing cards. On the game cards, there will be the word that the narrator student must explain to his group friends and five prohibited words right below this word. Prohibited words are synonyms, antonyms or close meanings of the word to be explained. According to the game rules, the student narrator will explain the word on the cards to his group friends without using prohibited words.
  Arms: Interversion group

SUMMARY:
Innovative learning methods can be used in teaching nursing history. One of the most preferred among these methods is learning through games. It is known that today's Generation Z students prefer active learning methods and want to learn by having fun instead of learning by rote. It is reported that learning through games improves students' knowledge and skills and increases retention. One of the methods of learning through games is the "tell me" game. The "Tell Me" game involves the narrator explaining the words prepared specifically for the subject to a group of students without using prohibited words. Other students in the group try to know the word explained. Thus, both the student narrator and the student trying to know actively use their critical thinking and decision-making skills. This research aims to determine the effect of the tell-all game used in teaching nursing history on students' learning and opinions.

DETAILED DESCRIPTION:
Nursing is a profession that emerged as a result of social needs and has very old roots. In order to evaluate the current situation of a profession, it is very important to know its history, the reasons for its emergence, the processes it has gone through from past to present, and its development processes. The contributions of the nursing profession to society and understanding its science and art dimensions can only be explained through the history of nursing. Therefore, the importance of professional history courses in nursing education cannot be denied. Teaching the history of nursing in detail strengthens the identity of nursing and develops students' critical thinking and problem-solving skills. It also allows nurses to demonstrate their self-efficacy. In addition, it helps develop a strong professional identity. In addition, improving nurses' historical knowledge directly affects their perception of the profession, attitude towards the profession, and nursing care. Correct historical awareness will enable nurses to learn from past practices and distinguish practices that are not suitable for nursing today. Therefore, it is very important to teach nursing history in undergraduate nursing education.The population of the research will consist of 200 second-year students enrolled in the Nursing History and Deontology course at the Faculty of Nursing of a state university in Turkey.Among the students who meet the criteria to participate in the research, 132 students will be determined by simple random sampling method by creating a simple random numbers table. The selected 132 students will be randomly assigned to two groups of 66 students (control and intervention) so that the overall academic achievement score of both groups is homogeneous.Data; It will be collected with the Introductory Features Form, Nursing History Knowledge Test and Nursing History Teaching Evaluation Form.

ELIGIBILITY:
Inclusion Criteria:

* Taking the nursing history and deontology course for the first time,
* Agreeing to participate in the research.

Exclusion Criteria:

* Graduating from a health-related high school or university,
* Having difficulty in speaking and understanding Turkish,
* Not participating in any of the research steps (theoretical training, explain game, topic repetition, pre-test, post-test),
* It means wanting to leave research.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Nursing History Knowledge Test | up to 4 months
  It will be used to determine students' knowledge of nursing history.

SECONDARY OUTCOMES:
Nursing History Teaching Evaluation Form | up to 4 months
  It will be used for students to evaluate nursing history teaching.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No